CLINICAL TRIAL: NCT07130604
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Phase III Study to Evaluate the Efficacy and Safety of D-2570 in Subjects With Moderate to Severe Plaque Psoriasis
Brief Title: Evaluate the Efficacy and Safety of D-2570 in Subjects With Moderate to Severe Plaque Psoriasis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: InventisBio Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D2570-301
Record Dates: First submitted 2025-08-12; First posted 2025-08-19 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Plaque Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- D-2570 group1 (Experimental)
  Interventions: Drug: D-2570
- D-2570 group2 (Experimental)
  Interventions: Drug: D-2570
- Placebo group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: D-2570 — Randomized in a 1:1:1 ratio through the randomization system, and assigned to D-2570 group1, group 2 or placebo group.
  Arms: D-2570 group1; D-2570 group2
Drug: Placebo — Randomized in a 1:1:1 ratio through the randomization system, and assigned to D-2570 group1, group 2 or placebo group.
  Arms: Placebo group

SUMMARY:
This study is a randomized, double-blind, placebo-controlled multicenter clinical trial targeting subjects with moderate to severe plaque psoriasis.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, placebo-controlled multicenter clinical trial targeting subjects with moderate to severe plaque psoriasis, with a total of 390 subjects planned to be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Subject voluntarily takes part in the study after being fully informed,signs a written ICF, and agrees to follow procedures specified in the study protocol;
2. Plaque psoriasis assessed by the investigator as suitable for systemic treatment and stable (defined as stable as no significant outbreak of morphological change or disease activity assessed by the investigator) for at least 6 months prior to signing informed consent;
3. During the screening period and before taking the investigational drug for the first time, psoriatic surface area (BSA) ≥10%, PGA score ≥ 3, PASI score ≥ 12;
4. Hematology, Blood chemistry and Urinalysis examination were basically normal.

Exclusion Criteria:

1. Erythrodermic psoriasis, pustular psoriasis, guttate psoriasis, reverse psoriasis, drug-induced psoriasis;
2. Have other skin lesions that affect the evaluation of treatment outcomes, such as eczema;
3. History of herpes zoster/herpes simplex, or presence of herpes zoster/herpes simplex infection during the screening period;
4. Have a history of tuberculosis, or active tuberculosis, or latent tuberculosis, or suspected clinical manifestations of tuberculosis infection;
5. Other conditions that the investigator considers inappropriate for participation in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Estimated)
Dates: Start 2025-09-18 (Actual); Primary Completion 2027-07-28 (Estimated); Study Completion 2027-07-28 (Estimated)

PRIMARY OUTCOMES:
The percentage of subjects with at least 90% improvement in PASI | Day 1-Day 112
  The percentage of subjects with at least 90% improvement in PASI from baseline at week 16 of treatment.

SECONDARY OUTCOMES:
Percentage of subjects with a PGA | Day 1-Day 112
  Percentage of subjects with a PGA score of 0 or 1 and ≥2 points from baseline at week 16 of treatment.
The percentage of subjects with at least 75% improvement in PASI | Day1-Day365
  The percentage of subjects with at least 75% improvement in PASI from baseline at each visit.
The percentage of subjects with at least 90% improvement in PASI | Day1-Day365
  The percentage of subjects with at least 90% improvement in PASI from baseline at each visit.
The percentage of subjects with at least 100% improvement in PASI | Day1-Day365
  The percentage of subjects with at least 100% improvement in PASI from baseline at each visit.
The percentage of subjects with improvement in PASI | Day1-Day365
  The percentage of subjects with improvement in PASI from baseline at each visit.
Percentage of subjects with a PGA | Day1-Day365
  Percentage of subjects with a PGA score of 0 or 1 and ≥2 points from baseline at each visit.
The percentage of subjects with at least 90% improvement in PASI | Day1-Day365
  The percentage of subjects with at least 90% improvement in PASI from baseline at week 16 of treatment and maintained response at Week 52.
Percentage of subjects with a PGA score of 0 or 1 and ≥2 points from baseline | Day1-Day365
  Percentage of subjects with a PGA score of 0 or 1 and ≥2 points from baseline at week 16 of treatment and maintained response at Week 52.
Percentage of subjects with baseline ss-PGA score ≥3 | Day 1-Day 112
  Percentage of subjects with baseline ss-PGA score ≥3 who achieved ss-PGA 0 or 1 at Week 16 of treatment.
Percentage of subjects with baseline PGA-F score ≥3 | Day 1-Day 112
  Percentage of subjects with baseline PGA-F score ≥3 who achieved ss-PGA 0 or 1 at Week 16 of treatment.
Percentage of subjects with baseline pp-PGA score ≥3 | Day 1-Day 112
  Percentage of subjects with baseline pp-PGA score ≥3 who achieved ss-PGA 0 or 1 at Week 16 of treatment.
Percentage of subjects with baseline DLQI score ≥2 | Day 1-Day 112
  Percentage of subjects with baseline DLQI score ≥2 who achieved DLQI 0 or 1 at Week 16 of treatment.
The main PK parameters -Time to maximum measured plasma concentration -Tmax Population pharmacokinetic characteristics of D-2570 | Day1-Day365
  The main PK parameters -Time to maximum measured plasma concentration -Tmax
The main PK parameters#Area under the plasma concentration versus time curve-AUC | Day1-Day365
  The main PK parameters#Area under the plasma concentration versus time curve-AUC
The main PK parameters-Vz/F (apparent volume of distribution) | Day1-Day365
  The main PK parameters-Vz/F (apparent volume of distribution)
The main PK parameters Half-life -t1/2 | Day1-Day365
  The main PK parameters Half-life -t1/2
The main PK parameters-CL/F (apparent clearance) | Day1-Day365
  The main PK parameters-CL/F (apparent clearance)
Weight and height will be combined to report BMI in kg/m^2 | Day1-Day365
  Weight and height will be combined to report BMI in kg/m^2
Incidence and severity of AEs based on NCI CTCAE V5.0 | Day1-Day365
  Incidence and severity of AEs based on NCI CTCAE V5.0
Incidence and severity of TEAEs based on NCI CTCAE V5.0 | Day1-Day365
  Incidence and severity of TEAEs based on NCI CTCAE V5.0

CONTACTS AND LOCATIONS:
Overall Officials: Jianzhong Zhang, Principal Investigator — Study Official is required by the WHO and ICMJE.
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No